CLINICAL TRIAL: NCT07043816
Title: Impact of PharmaTE Trial on Glycemic Control, Diabetes Knowledge, Medication Adherence and Quality of Life in Type 2 Diabetes Patients: A Mixed-Method Study Protocol
Acronym: PharmaTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabia Hussain (Other)
Collaborators: Universiti Sains Malaysia (Other)
Responsible Party: Sponsor-Investigator, Rabia Hussain, DR. Rabia Hussain, Principal Investigator, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: USM-DSAP-2025-002
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes (T2DM); Glycemic Control; Diabetes Knowledge; Medication Adherence; Quality of Life
Keywords: PharmaTE
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention study, the clinical pharmacist conducting the PharmaTE trial will be aware of whether the patient will be assigned to the PharmaTE trial interventional group (IG) or control (non-blinded). However, the investigators who will collect the data from each patient before and after the intervention will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients randomized to the control group will receive standard care provided in a diabetes excellence center, including nurse assessment, physician assessment, and care provision by a multidisciplinary team. They will also visit the hospital pharmacy to fill their prescriptions without further clinical pharmacist intervention. However, there will be no restriction on contacting the clinical pharmacist for advice.
- Interventional Group (PharmaTE group) (Experimental): In addition to standard care, patients in the PharmaTE trial interventional group will receive tele-education led by a clinical pharmacist who has completed a training course and is certified as a diabetes educator. The tele-education program is comprised of five individualized educational sessions, each lasting approximately 20-30minutes and held at two-month intervals. These sessions are conducted via Zoom or telephone based on patient preference. Before the beginning of each session, participants will receive a reminder message along with the Zoom meeting invitation link about the session, covering various educational topics related to diabetes management. Additionally, after each session, patients will receive a brochure summarizing what has been discussed.
  Interventions: Behavioral: PharmaTE Trial

INTERVENTIONS:
Behavioral: PharmaTE Trial — In addition to standard care, patients in the PharmaTE trial interventional group will receive tele-education led by a clinical pharmacist who has completed a training course and is certified as a diabetes educator. The tele-education program is comprised of five individualized educational sessions, each lasting approximately 20-30minutes and held at two-month intervals. These sessions are conducted via Zoom or telephone based on patient preference. Before the beginning of each session, participants will receive a reminder message along with the Zoom meeting invitation link about the session, covering various educational topics related to diabetes management. Additionally, after each session, patients will receive a brochure summarizing what has been discussed.
  Arms: Interventional Group (PharmaTE group)

SUMMARY:
The goal of this clinical trial is to find out whether a pharmacist-led tele-educational program (PharmaTE trial) can help people with type 2 diabetes manage their condition better.

The main questions this study aims to answer are:

1. Does the PharmaTE trial improve blood sugar control (HbA1c levels)?
2. Does it help patients better understand their condition?
3. Does it increase how well patients follow their medication schedule?
4. Does it improve the quality of life for patients with type 2 diabetes?
5. Is this type of tele-education program feasible and acceptable for patients?

Participants will:

Be randomly placed into one of two groups:

Intervention group: Receive five virtual education sessions with a clinical pharmacist over the phone or via Zoom (each lasting 20-30 minutes), in addition to their usual diabetes care.

Control group: Continue receiving standard diabetes care from their healthcare team without the additional pharmacist-led sessions.

Complete assessments at the beginning and end of the study. These include:

A blood test for HbA1c

, Questionnaires on diabetes knowledge, medication adherence, and quality of life

Some participants in the intervention group will be invited for interviews after the sessions to share their experiences and opinions about the program.

Who can join? Adults aged 18-65 with uncontrolled type 2 diabetes (HbA1c > 7%), receiving care at Ibrahim Bin Hamad Obaidullah Hospital in Ras Al-Khaimah, who speak Arabic and can provide consent.

DETAILED DESCRIPTION:
This study evaluates the impact of a clinical pharmacist-led tele-educational intervention (PharmaTE trial) on glycemic control, diabetes knowledge, medication adherence, and quality of life among adult patients with type 2 diabetes mellitus (T2DM) at a secondary care hospital in Ras Al Khaimah, United Arab Emirates.

The rationale for the study stems from the increasing prevalence of T2DM in the region, with many patients experiencing poor glycemic control and limited access to diabetes education. Previous evidence suggests that pharmacist-led interventions can improve treatment adherence and health outcomes. However, such approaches, particularly via tele-education, remain underexplored in the UAE healthcare setting.

This is a mixed-methods study with an embedded design consisting of a prospective, randomized controlled trial (RCT) and a qualitative component. A total of 154 eligible adult patients with uncontrolled T2DM (HbA1c > 7%) will be randomly assigned to either an intervention group or a control group. The intervention group will receive five tele-education sessions delivered by a clinical pharmacist, focusing on key aspects of diabetes self-management. The control group will continue to receive standard care without pharmacist-led education.

Baseline and post-intervention assessments (after 3 months) will include HbA1c levels, patient knowledge (Michigan Diabetes Knowledge Tool), medication adherence (MMAS-8), and quality of life (DQoL). A subset of intervention participants will also be interviewed to explore the feasibility and acceptability of the program.

The findings are expected to support the integration of pharmacists into diabetes care models and inform future digital health strategies.

ELIGIBILITY:
Inclusion Criteria

* Patients diagnosed with uncontrolled type 2 diabetes (defined as glycated haemoglobin [HbA1c] >7%) within the previous 12 months
* Adults (18 to 65 years) of either gender
* Prescribed at least one antidiabetic medication
* Have access to either a telephone or a mobile phone
* Treated in an outpatient facility in IBOH, RAK
* Arabic-speaking patients
* Patients who understand study information and are given written informed consent.

Exclusion Criteria:

* Under 18 years old
* Pregnant ladies
* Patients admitted to the emergency department
* Patients with severe hepatic or renal dysfunction
* Diagnosed with type 1 DM or diagnosed with gestational diabetes
* Having vision or hearing impairments and psychological problems
* Immunocompromised patients, e.g., organ transplants, AIDS, cancer patients, and patients on immunosuppressant therapy
* Patients with no or limited access to either a telephone or mobile phone, as well as those without reliable internet access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control | Both groups will assessed at baseline and after the end of the intervention (3 months after completing the intervention). Patients whose has been measured within the last two weeks will not be required to undergo repeat testing.
  The primary outcome is improved glycemic control compared to the baseline. The glycemic level will be assessed evaluating the HbA1c level at baseline and after intervention completion in both the interventional and control group Glycemic levels are considered normal when HbA1c level is within predefined ranges as suggested by the America Diabetes Association (ADA), which recommends that adults with diabetes maintain an HbA1c of less than 6.5 % (Eet al., 2024, 2025).

SECONDARY OUTCOMES:
Diabetes Knowledge | Both groups will assessed at baseline and after the end of the intervention (3 months after completing the intervention).
  Patient knowledge about diabetes will be assessed using the Michigan Diabetes Knowledge Test (MDKT), which is validated tool that has been utilized in several settings to evaluate diabetic patients' knowledge. The Michigan survey instruments have been translated into several languages (Collins et al., 2011; Fitzgerald et al., 2016). The Michigan Knowledge Test (MDKT) is comprised of 14 multiple-choice questions. The knowledge test scores ranged from 0 to 14 with 14 representing the highest level of knowledge of diabetes and zero representing the lowest. We considered the knowledge score of <7 constituted poor knowledge, 7-11 moderate knowledge, and 12-14 good knowledge (Al-Aal., 2016). The Arabic version of the MDKT will be utilized, and permission for its use has been obtained from the to developer (Alhaiti et al., 2016).
3. Medication Adherence | Both groups will assessed at baseline and after the end of the intervention (3 months after completing the intervention).
  Medication Adherence will be assessed to evaluate the patient's compliance with their treatment regimen using the Arabic version of Morisky Medication Adherence Scale (MMAS-8), The MMAS-8 is a validated assessment tool developed by Morisky et al (Morisky et al., 1986). MMAS-8 has good validity and reliability, has also been proven to be a useful screening technique for chronic disease medications, and has been validated on other Arabic patients suffering from chronic diseases (W.-Y. Lee et al., 2013; Sweileh et al., 2014).
Diabetic Quality of Life | Both groups will assessed at baseline and after the end of the intervention (3 months after completing the intervention).
  The Diabetes Quality of Life (DQoL) questionnaire will assess diabetes quality of life (Al-Qerem et al., 2021). The questionnaire consists of 29 items divided into three factors: Satisfaction (14 items), Impact (11 items), and Worries (4 items). The satisfaction and impact questions include a 5-point Likert scale [very satisfied (1 point), quite satisfied, satisfied, little satisfied, and very dissatisfied (5 points)].
  The DQOL questionnaire has been previously field-tested and validated for its administration in type 2 diabetic patients and shown to be internally consistent, reproducible, and responsive. It is commonly used and translated into several languages, including Arabic. The Arabic version of the DQOL questionnaire has previously been validated.

OTHER OUTCOMES:
Feasibility and Acceptability | Three months after completing the intervention
  After completing the quantitative assessments, a semi-structured interview will be conducted with a subset of patients from the intervention group, three months after the intervention, via either a virtual meeting or a phone call, based on their preference. The interviews will focus on participants' feedback, challenges faced, and perceptions of the intervention's feasibility and acceptability. Semi-structured interviews will be conducted using an interview guide. With participants' consent, interviews will be audio-recorded, and then will be transcribed verbatum.
  A purposive sampling technique will be used for recruiting the patients, the sample size is guided by data saturation for qualitative research, whereby no new themes appear from the data (Glaser & Strauss, 2017) It is anticipated that 15 to 25 interviews will be required to achieve data saturation (Glaser & Strauss, 2017).

IPD SHARING:
Plan to Share IPD: Undecided